CLINICAL TRIAL: NCT05855603
Title: Recurrent Cardioinhibitory Reflex Syncope. PermANent PAcemaker Therapy or CardionEuroablation? A Multicenter RAndomized Clinical Trial
Brief Title: Cardioinhibitory Reflex Syncope. Permanent Pacemaker Therapy or Cardioneuroablation?
Acronym: PANACEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Rodolfo San Antonio, Medical Doctor, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICPS044/22
Record Dates: First submitted 2023-04-20; First posted 2023-05-11 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Reflex Syncope
Keywords: Cardioneuroablation; Permanent cardiac pacing; Vasovagal syncope
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardioneuroablation (Experimental): Bi-atrial ablation of GPs: CARDIONEUROABLATION (Group A, n = 45)
  Interventions: Procedure: Cardioneuroablation
- Dual-chamber pacemaker (Active Comparator): Implant of a dual-chamber CLS PACEMAKER* (Group B, n = 45).
  *or failing this, a dual-chamber pacemaker with RDR algorithm
  Interventions: Device: Permanent pacemaker therapy

INTERVENTIONS:
Procedure: Cardioneuroablation — Ganglionated plexi will be localized using an empirical anatomical approach and/or a fractionated electrogram-based strategy.
  Point-by-point ablation will be performed using radiofrequency energy and an irrigated tip contact force sensing ablation catheter in a power control mode (35-50 W; AI, 350-500; LSI, 4.5-5.5). The right superior GP (RSGP), left superior GP (LSGP) and posterior left GP (PMLGP) will be targeted during CNA. Radiofrequency applications in other GPs will be left at the discretion of the operator.
  At the end of the procedure, another EP study and atropine test will be performed. Clinical endpoints for completion of the CNA will be: 1) a HR increase >20% if the CNA was performed under general anesthesia/deep sedation; 2) improved electrophysiological parameters; 3) significant reduction in atropine response (HR increase <10% after atropine); and 4) in case of using extracardiac vagal stimulation, lack of response.
  Arms: Cardioneuroablation
Device: Permanent pacemaker therapy — All patients in the pacemaker group will receive a dual-chamber pacemaker that has the ability to be programmed in the DDD-CLS algorithm mode (or failing this, a dual-chamber pacemaker with RDR algorithm).
  Arms: Dual-chamber pacemaker

SUMMARY:
Reflex syncope is the most common form of syncope. It can lead to injuries and affect quality of life. Nonpharmacological and medical therapies have limited effectiveness. In certain patients, cardiac pacing seem to be beneficial. More recently cardioneuroablation (CNA) has emerged as a novel therapy for reflex syncope. The investigators aim to determine whether CNA is more effective than cardiac pacing at reducing the rate of cardioinhibitory-type reflex syncope.

DETAILED DESCRIPTION:
Reflex or neurally mediated syncope is the most common form of syncope in any setting and at all ages. It is associated with an autonomic imbalance in which vagal hyperactivity predominates, resulting in vasodilation or bradycardia or both, thereby producing a fall in global cerebral perfusion. It is divided into three types: vasovagal, situational, and carotid sinus syndrome.

Reflex syncope is benign and usually occurs in healthy people; however, very frequent syncope or events without prodromal symptoms can lead to injuries and affect long-term quality of life. Nonpharmacological and medical therapies proven effective in randomized clinical trials are scarce. In certain patients with frequent and burdensome cardioinhibitory reflex syncope, dual-chamber cardiac pacemakers seem to be beneficial. More recently, catheter-based cardiac autonomic modulation, or cardioneuroablation (CNA), has emerged as a novel therapy for reflex syncope, and positive results in small open-label cohort studies, and more recently in the first randomized study, have been reported.

The literature provides sufficient evidence that cardiac pacing should be considered in select patients affected by severe forms of reflex syncope with frequent recurrence and a high risk of injury. Current guidelines suggest that pacemaker therapy should be considered in patients aged more than 40 years with frequent recurrent reflex syncope when asystole has been documented, induced by either carotid sinus massage (CSM) or the head-up tilt test (HUTT), or recorded using an electrocardiogram (ECG) monitoring system (≥3 seconds if syncope, ≥6 seconds if asymptomatic).

Cardiac autonomic system modulation by endocardial ablation targeting atrial ganglionated plexi (GPs), or CNA, has been recently proposed as a novel therapy for reflex syncope.

Cardioneuroablation was introduced by Pachon et al. in 2005. In their initial study, twenty-one symptomatic patients with vasovagal syncope (6 patients), functional high-degree atrio-ventricular block (7 patients), and/or functional sinus node dysfunction (13 patients), were treated with CNA without complications. Follow-up for a mean of 9.2 months demonstrated symptom relief for all patients. After this initial description, several small studies and case series confirmed the efficacy of this approach. In a recent randomized prospective study, Piotrowski et al. documented that not only could CNA significantly reduce recurrences of syncopal episodes in patients with vasovagal syncope, it could also improve quality of life.

The primary strength of this therapeutic approach is that it avoids pacemaker implant, a procedure with a significant complication rate during long-term follow-up in a population composed predominantly of young and otherwise healthy patients.

The excellent results reproduced by many investigators worldwide suggest that CNA should be considered in patients with reflex syncope, especially those who display an important cardioinhibitory component of syncope. However, given that current evidence is limited, and the procedure carries potential risk, a randomized clinical trial to assess the true benefit of CNA and to compare this technique with pacemaker implantation should be performed. Results could guide the physician to the best current choice in this scenario.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 40 years.
* Having a 12-month history that includes at least two documented episodes of spontaneous reflex syncope or one episode that led to injury in addition to at least two presyncopal events, refractory to all recommended types of standard treatment.
* Bradycardia-syncope correlation (at least 3 seconds of asystole due to sinus arrest or atrio-ventricular block) confirmed by ECG during spontaneous syncope.
* If lacking ECG evidence during spontaneous syncope, a cardioinhibitory response (VASIS type 2A or 2B) on tilt test.
* Displaying indicators for pacing such as those suggested in the ESC guidelines for a class I recommendation for patients with reflex syncope.
* Significantly decreased quality of life due to syncope.
* Sinus rhythm on ECGs.
* Obtained written informed consent.

Exclusion Criteria:

* Intrinsic sinus or atrioventricular nodal disease with a proven indication for permanent pacemaker implantation.
* Evidence of structural heart disease.
* Contraindications to ablation in the right or left atrium.
* Life expectancy <12 months.
* Lacking willingness to comply with the randomization procedure.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of CNA in the treatment of cardioinhibitory reflex syncope in comparison to pacemaker therapy. | 12 months
  Differences in 12-month syncope-free survival between the 2 groups

SECONDARY OUTCOMES:
To evaluate the incidence of complications in the short and long terms for CNA compared to pacemaker therapy | 1 and 12 months
  Pacemaker and CNA complication rates at 1 and 12 months
In patients undergoing CNA, evaluation of the degree of long-term reinnervation using the tilt table test (HUTT) | 1 and 12 months
  Changes in response to HUTT (type 1-3) at baseline, 1 and 12 months
In patients undergoing CNA, evaluation of the degree of long-term reinnervation using the atropine test | 1 and 12 months
  Changes in response (maximum heart rate) to atropine test at baseline, 1 and 12 months
To determine which of the 2 strategies, CNA or cardiac pacing, is superior at preventing a composite of syncope and presyncope | 12 months
  Differences in 12-month syncope- and presyncope-free survival between the 2 groups
Evaluations of changes in quality of life, comparing the two therapies | 12 months
  Using the Impact of Syncope on Quality-of-life questionnaire (University of Calgary). It consists of 9 questions with 6 choices and 3 questions with 5 choices. The overall maximum score is 57. The higher the score, the poorer the QOL is
To determine if CNA produces variations in the QTc interval | 12 months
  The QTc interval will be measured at minimum, average and maximum heart rate using a 24-hour holter monitoring
To determine if CNA produces variations in the burden of atrial or ventricular arrhythmias compared to pacemaker therapy | 12 months
  Arrhythmias will be detected by implantable loop recorder in the group A (CNA) vs. by the pacemaker itself in group B

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo San Antonio, MD, PhD, Study Chair — Hospital Universitario de Bellvitge
Locations (10):
- Spain (10):
  - Hospital Universitario San Juan de Alicante, Sant Joan d'Alacant, Alicante
  - Hospital Universitari General de Castellón, Castellon, Castellón
  - Hospital Universitario Álvaro Cunqueiro de Vigo, Vigo, Pontevedra
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276
- [Result] Aksu T, Gupta D, D'Avila A, Morillo CA. Cardioneuroablation for vasovagal syncope and atrioventricular block: A step-by-step guide. J Cardiovasc Electrophysiol. 2022 Oct;33(10):2205-2212. doi: 10.1111/jce.15480. Epub 2022 Apr 9. PMID 35362165
- [Result] Piotrowski R, Baran J, Sikorska A, Krynski T, Kulakowski P. Cardioneuroablation for Reflex Syncope: Efficacy and Effects on Autonomic Cardiac Regulation-A Prospective Randomized Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):85-95. doi: 10.1016/j.jacep.2022.08.011. Epub 2022 Aug 28. PMID 36114133